CLINICAL TRIAL: NCT03891355
Title: Carfilzomib (K) Plus Lenalidomide (R) and Dexamethasone (D) for BTK Inhibitors Relapsed-refractory or Intolerant Mantle Cell Lymphomas: a Phase II Study
Brief Title: Carfilzomib + Lenalidomide and Dexamethasone for BTK Inhibitors Relapsed-refractory or Intolerant MCL
Acronym: FIL_KLIMT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fondazione Italiana Linfomi - ETS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FIL_KLIMT
Record Dates: First submitted 2019-03-15; First posted 2019-03-27 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Mantle Cell Lymphoma
Keywords: Carfilzomib; Lenalidomide; Dexamethasone; relapsed-refractory or intolerant mantle cell lymphomas
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — carfilzomib; Lenalidomide; Dexamethasone

STUDY DESIGN:
Intervention Model Description: This is a prospective, multicenter, single arm, phase II trial designed to evaluate the safety and efficacy of the combination of Carfilzomib (K), Lenalidomide (R) and Dexamethasone (D) in patients with mantle cell lymphoma (MCL) relapsed/refractory (R/R) or intolerant to BTK inhibitor (BTKi) monotherapy or BTKi containing regimens.
  The primary endpoint will be assessed 12 months after the start of treatment of the last patient. However, responsive patients (CR, PR, SD) may continue to receive K up to a maximum of 24 cycles and RD up to a maximum of 24 cycles. Patients who will interrupt therapy (for any reason) will be followed up to 12 months after the end of the treatment.
  After checking inclusion and exclusion criteria and signing written informed consent, the patient will be enrolled with an identification numeric code.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Carfilzomib (K) plus Lenalidomide (R) and Dexamethasone (D) (Experimental): Carfilzomib (K) (maximum period of treatment= 24 cycles)
  * K on days 1-2, 8-9, 15-16 during cycles 1-12. The dosage of K will be 20 mg/m2 10' iv infusion on day 1 and 2 during cycle 1 and then 27 mg/m2 10' iv infusion thereafter;
  * K: on days 1-2, 15-16 during cycles 13-24. The dosage of K will be 27 mg/m2 10' iv infusion. Lenalidomide (R) (maximum period of treatment= 24 cycles)
  * R: 25 mg/daily on day 1 to 21 of a 28 days course; for patients with creatinine clearance ≥ 30 mL/min but < 50 mL/min the dosage of R will be 10 mg/daily on day 1 to 21 of a 28 days course.
  Dexamethasone (D) (maximum period of treatment= 24 cycles) PO or IV D on days 1-2, 8-9, 15-16, 22-23. The dosage will be 20 mg between 30 minutes and 4 hours prior to K. For patients older than 75 years the dosage may be reduced at 10 mg.
  Interventions: Drug: Carfilzomib; Drug: Lenalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Carfilzomib — Carfilzomib
Drug: Lenalidomide — Lenalidomide
Drug: Dexamethasone — Dexamethasone

SUMMARY:
This is a prospective, multicenter, single arm, phase II trial designed to evaluate activity and the safety of the combination of Carfilzomib (K), Lenalidomide (R) and Dexamethasone (D) in patients with mantle cell lymphoma (MCL) relapsed/refractory (R/R) or intolerant to BTK inhibitor (BTKi) monotherapy or BTKi containing regimens with active disease necessitating treatment.

DETAILED DESCRIPTION:
This is a prospective, multicenter, single arm, phase II trial designed to evaluate the safety and efficacy of the combination of Carfilzomib (K), Lenalidomide (R) and Dexamethasone (D) in patients with mantle cell lymphoma (MCL) relapsed/refractory (R/R) or intolerant to BTK inhibitor (BTKi) monotherapy or BTKi containing regimens.

The primary endpoint will be assessed 12 months after the start of treatment of the last patient. However, responsive patients (CR, PR, SD) may continue to receive K up to a maximum of 24 cycles and RD up to a maximum of 24 cycles. Patients who will interrupt therapy (for any reason) will be followed up to 12 months after the end of the treatment.

ELIGIBILITY:
Inclusion criteria Patient has a confirmed diagnosis of MCL according to the WHO 2017 classification;

* Previous treatment with BTKi monotherapy or BTKi containing regimens with R/R disease; and/or patients who discontinued BTKi monotherapy or BTKi containing regimens for adverse events and have active disease necessitating treatment;
* Previous treatment with Lenalidomide is accepted if patient resulted responsive and interrupted Lenalidomide at least 12 months before enrollment to this study;
* Patient age is ≥ 18 < 80 years;
* Patient has an Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2;
* Understands and voluntarily signs an informed consent form;
* Able to adhere to the study visit schedule and other protocol requirements; Patient has at least one site of measurable nodal disease at baseline ≥ 2.0 cm in the longest transverse diameter as determined by CT scan (MRI is allowed only if CT scan cannot be performed). Note: Patients with bone marrow involvement are eligible;
* Adequate hematological counts: ANC > 1.5 x 109/L and platelet count > 75 x 109/L unless due to bone marrow involvement by MCL;
* Conjugated bilirubin up to 2 x ULN unless due to liver involvement by MCL;
* Alkaline phosphatase and transaminases up to 2 x ULN unless due to liver involvement by MCL;
* Creatinine clearance ≥ 30 ml/min; a dose reduction of Lenalidomide for patients with creatinine clearance ≥ 30 mL/min but < 50 mL/min is planned;
* Patient has the ability to swallow capsules or tablets;
* Life expectancy ≥ 2 months;
* Male and Female patients: accordance to comply with Lenalidomide Risk Management Plan for pregnancy prevention.

Exclusion criteria

* Patient who have received an experimental drug or used an experimental medical device within 4 weeks before the planned start of treatment. Concurrent participation in non-treatment studies is allowed, if it will not interfere with participation in this study;
* Patient has a history of CNS involvement with lymphoma;
* Patient with previous history of malignancies (apart MCL) ≤ 3 years before study accrual with the exception of currently treated basal cell and squamous cell carcinoma of the skin, or carcinoma "in situ" of the cervix;
* History of clinically relevant liver or renal insufficiency; significant cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, rheumatologic, hematologic, psychiatric, or metabolic disturbances;
* Patient has any other concurrent severe and/or uncontrolled medical condition(s) (e.g., uncontrolled diabetes mellitus, uncontrolled hypertension, active/symptomatic coronary artery disease, chronic obstructive pulmonary disease (COPD), active hemorrhage, psychiatric illness, active or uncontrolled infection that in the investigator opinion places the patient at unacceptable risk and would prevent the subject from signing the informed consent form;
* Creatinine clearance < 30 ml/min;
* Significant neuropathy (Grades 3 - 4, or Grade 2 with pain) within 14 days prior to enrollment;
* Known history of allergy to Captisol® (a cyclodextrin derivative used to solubilize Carfilzomib);
* Contraindication to any of the required concomitant drugs or supportive treatments or intolerance to hydration due to preexisting pulmonary or cardiac impairment;
* Patients with LVEF <40%
* Patients with New York Health Association (NYHA) Class III and IV heart failure; myocardial infarction in the preceding 6 months; conduction abnormalities, including but not limited to atrial fibrillation, atrioventricular (AV) block, QT prolongation, sick sinus syndrome, ventricular tachycardia;
* Patients with severe bradycardia (heart rate <40 bpm, hypotension, light-headedness, syncope);
* Acute active infection requiring treatment (systemic antibiotics, antivirals, or antifungals) within 14 days prior to enrollment;
* Patients with active pulmonary embolism or deep vein thrombosis (diagnosed within 30 days of study enrollment);
* Patient has a known history of HIV seropositivity;
* Patient has active HBV hepatitis. The following categories of HBV positive patients but with no evidence of active hepatitis may be considered for the study:

  * patient is HBsAg + with HBV DNA < 2000 UI/ml (inactive carriers); HBV DNA > 2000 UI/ml is criteria of exclusion;
  * patient is HBsAg - HBsAb +;
  * patient is HBsAg - but HBcAb +
* Patient with HCV active hepatitis are excluded from the study. Patient with no evidence of active hepatitis and/or advanced chronic liver disease according to liver biopsy or fibro-scan evaluation may be included into the study;
* Previous treatment with Lenalidomide if patient resulted primary refractory to Lenalidomide or interrupted Lenalidomide less than 12 months before enrollment to this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2020-12-04 (Actual); Study Completion 2022-12-08 (Estimated)

PRIMARY OUTCOMES:
Primary Efficacy Endpoint - 12-months overall survival | The primary endpoint will be assessed 12 months after the start of treatment of the last patient.
  12-month overall survival : probability of surviving from the date of beginning of therapy up to month 12 based on Kaplan-Meier estimator

SECONDARY OUTCOMES:
Secondary Endpoints 1 - ORR | The endpoint will be assessed from the date of randomization to the date of the first documented progression, evaluated up to 12 months.
  overall response rate will be defined according to Lugano criteria. The best overall
  response will be defined as the best response between the date of beginning of therapy and the last restaging. Patients without response assessment (due to whatever reason) will be considered as non-responders.
Secondary Endpoints 1 - CR | The endpoint will be assessed from the date of randomization to the date of the first documented progression, evaluated up to 12 months.
  complete response rate between the date of beginning of therapy and the last restaging. Patients without response assessment (due to whatever reason) will be considered as non-responders.
Secondary Endpoints 1 - PR | The endpoint will be assessed from the date of randomization to the date of the first documented progression, evaluated up to 12 months.
  partial response rate between the date of beginning of therapy and the last restaging. Patients without response assessment (due to whatever reason) will be considered as non-responders.
Secondary Endpoints 1 - SD | The endpoint will be assessed from the date of randomization to the date of the first documented progression, evaluated up to 12 months.
  rate between the date of beginning of therapy and the last restaging. Patients without response assessment (due to whatever reason) will be considered as non-responders.
Secondary Endpoints 2 - PFS | The endpoint will be assessed from the date of randomization to the date of the first documented progression, evaluated up to 12 months.
  progression-free survival will be defined as the time from beginning of therapy until lymphoma relapse or progression or death as a result of any cause; responding patients and patients who are lost to follow up will be censored at their last assessment date;
Secondary Endpoints 3 - OS | through the completion of the study, an average of 1 year
  overall survival will be defined as the time from beginning of therapy until death as a result of any cause; patients who are lost to follow up will be censored at their last assessment date;
Secondary Endpoints 4 - TTR | through the completion of the study, an average of 1 year
  time to response will be defined for all patients who achieved a response (Complete Response or Partial Response) and is measured from the date of beginning of therapy until the date of response. Patients in relapse or progression will be censored at their last assessment date. Patients death due to any cause will be consider censored or competing event according to different analysis plan
Secondary Endpoints 5 - DoT | through the completion of the study, an average of 1 year
  the duration of the treatment will be defined as the time from beginning of therapy until discontinuation due to any reason.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Zaja, Prof., Principal Investigator — Ospedale Maggiore Azienda Sanitaria Universitaria Trieste Ematologia
Locations (11):
- Italy (11):
  - ASST Spedali Civili di Brescia - Ematologia, Brescia
  - Fondazione IRCCS Istituto Nazionale dei Tumori di Milano - Ematologia, Milan
  - ASST Grande Ospedale Metropolitano Niguarda - SC Ematologia, Milan
  - AOU Maggiore della Carità di Novara - SCDU Ematologia, Novara
  - IRCCS Policlinico S. Matteo di Pavia - Div. di Ematologia, Pavia
  - Ospedale delle Croci - Ematologia, Ravenna
  - AOU Senese - U.O.C. Ematologia, Siena
  - A.O.U. Citta della Salute e della Scienza di Torino - Ematologia Universitaria, Torino
  - Azienda sanitaria-universitaria integrata Trieste (ASUITS) - SC Ematologia, Trieste
  - Azienda Sanitaria Universitaria Integrata di Udine (A.S.U.I. Udine) - SOC Clinica Ematologica, Udine
  - AOU Integrata di Verona - U.O. Ematologia, Verona

IPD SHARING:
Plan to Share IPD: No